CLINICAL TRIAL: NCT05326230
Title: A Clinical Study of the Ultrasound Renal Denervation System (PRDS-001) in Patients With Hypertension
Brief Title: A Clinical Study of the Paradise™ Renal Denervation System in Patients With Hypertension (RADIANCE-HTN DUO)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Otsuka Medical Devices Co., Ltd. Japan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDN-21-002
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Hypertension; Vascular Diseases; Cardiovascular Diseases
Keywords: Denervation; Hypertension
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Renal Denervation (Experimental): Renal Angiogram and Renal Denervation (PRDS-001- Paradise™ System)
  Interventions: Device: Paradise™ (PRDS-001) Renal Denervation Ultrasound System
- Sham Control (Sham Comparator): Renal Angiogram
  Interventions: Device: Renal Angiogram

INTERVENTIONS:
Device: Paradise™ (PRDS-001) Renal Denervation Ultrasound System — Following renal angiogram according to standard procedures, subjects remain blinded and are randomized to treatment with renal denervation or sham control
  Other Names: Renal Angiogram/Renal Denervation
  Arms: Renal Denervation
Device: Renal Angiogram — Following renal angiogram according to standard procedures, subjects remain blinded and renal angiogram is considered the sham procedure
  Arms: Sham Control

SUMMARY:
To compare the antihypertensive effect of renal denervation with the Paradise™ system with that of a sham procedure in hypertensive patients receiving two antihypertensive drugs at the time of consent, and treated with a duo combination antihypertensive pill.

ELIGIBILITY:
Inclusion Criteria :

* Patients who have received antihypertensive treatment with two antihypertensive drugs (ARB/ACE inhibitor and Ca channel antagonist, either as a single agent or as a combination) for at least 4 weeks prior to obtaining consent, with no change in the type or dosage.
* Patients with a mean seated office blood pressure of between 140 mmHg and 180 mmHg systolic and between 90 mmHg and 110 mmHg diastolic at screening visit.
* Patients with a mean 24-hour ABPM (ambulatory blood pressure measurement) of between 130 mmHg and 170 mmHg systolic and between 80 mmHg and 105 mmHg diastolic at baseline visit

Exclusion Criteria

* Lacks appropriate renal artery anatomy for renal denervation
* Secondary hypertension other than sleep apnea
* Type 1 diabetes mellitus or uncontrolled Type 2 diabetes
* Any history of cerebrovascular event or severe cardiovascular event, within 6 months prior to consent
* Repeated hospitalization for hypertensive crisis (twice or more) within 12 months prior to obtaining consent, or any hospitalization for hypertensive crisis within 3 months prior to obtaining consent
* Patients prescribed to drugs that have antihypertensive effects for other chronic diseases, and the investigator considers that discontinuation of these drugs may pose a serious risk to health
* Patients who are taking drugs known to affect blood pressure and the investigator judges that it is not possible to discontinue these drugs during the study period
* Patients with a history of persistent or permanent atrial tachyarrhythmia
* Patients with active implantable medical devices
* Primary pulmonary hypertension
* Patients with contraindications or unacceptable anaphylactic reactions or uncontrolled allergy to contrast media
* Night shift workers
* Pregnant, nursing or planning to become pregnant
* Patients with any of the following central laboratory tests at screening

  * Plasma aldosterone/renin ratio greater than or equal to 200 and plasma aldosterone greater than or equal to 60 pg/ml
  * HbA1c greater than or equal to 8.0%
  * eGFR less than 40 mL/min/1.73m2

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Mean change in 24-hour systolic ABPM | From baseline to 3 months post-procedure

SECONDARY OUTCOMES:
Mean change in 24-hour systolic ABPM | from baseline to 6 months post-procedure
Mean change in daytime/nighttime /24-hour ABPM (systolic/diastolic) (excluding primary and important secondary endpoints) | From baseline to 3, 6, 12 months post-procedure
Change in mean sitting office blood pressure (systolic/diastolic) | From baseline to 1, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 60 months post-procedure
Change in mean home blood pressure (systolic/diastolic) | From baseline to 1, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 60 months post-procedure
Percentage of subjects with a mean decrease in daytime/nighttime/24-hour systolic ABPM of ≥5 mmHg, ≥10 mmHg, and ≥15 mmHg | 3, 6, and 12months post-procedure
Percentage of subjects who required a change in antihypertensive medication | at any time up to 12 months after the procedure
Percentage of subjects who achieved blood pressure control without any change in antihypertensive medication | 3, 6, 12 months after the procedure
Percentage of subjects whose blood pressure was controlled by changing antihypertensive medication | 3, 6, 12 months after the procedure
Change in mean pulse pressure (difference between systolic and diastolic blood pressure) in the office, home, ABPM | 3, 6, 12 months after the procedure
Change in mean heart rate in the office, home, ABPM | 3, 6, 12 months after the procedure

CONTACTS AND LOCATIONS:
Locations (51):
- Japan (51):
  - Hirosaki University Hospital, Hirosaki-shi, Aomori
  - Tokyo Bay Urayasu Ichikawa Medical Center, Urayasu-shi, Chiba
  - Ehime University Hospital, Toon-shi, Ehime
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Fukuoka Sanno Hospital, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Iwaki City Medical Center, Iwaki, Fukushima
  - Chuno Kousei Hospital, Seki-shi, Gifu
  - Hiroshima City North Medical Center Asa Citizens Hospital, Hiroshima, Hiroshima
  - Nayoro City General Hospital, Nayoro-shi, Hokkaido
  - Sapporo-Kosei General Hospital, Sapporo, Hokkaido
  - Tonan Hospital, Sapporo, Hokkaido
  - Tomakomai City Hospital, Tomakomai-shi, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Nishinomiya Municipal Central Hospital, Nishinomiya-Shi, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Saiseikai Yokohamashi Nanbu Hospital, Yokohama, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Yokohama Rosai Hospital, Yokohama, Kanagawa
  - Chikamori Hospital, Kochi, Kochi
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Suzuka Chuo General Hospital, Suzuka-Shi, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - Niigata City General Hospital, Niigata, Niigata
  - Okayama Rosai Hospital, Okayama, Okayama-ken
  - Ryukyu University Hospital, Naha, Okinawa
  - Osaka Saiseikai Nakatsu Hospital, Osaka, Osaka
  - Osaka Rosai Hospital, Sakai-shi, Osaka
  - National Cerebral and Cardiovascular Center, Suita-shi, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Imamura Hospital, Tosu-shi, Saga-ken
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - Mitsui Memorial Hospital, Chiyoda-ku, Tokyo
  - St. Luke's International Hospital, Cyuo-ku, Tokyo
  - Minamino Junkanki Hospital, Hachioji-shi, Tokyo
  - Kimura Clinic, Meguro-Ku, Tokyo
  - Toho University Medical Center Ohashi Hospital, Meguro-ku, Tokyo
  - Tokyo Saiseikai Central Hospital, Minato-ku, Tokyo
  - Tokyo Takanawa Hospital, Minato-ku, Tokyo
  - Toranomon Hospital, Minato-ku, Tokyo
  - Japanese Red Cross Musashino Hospital, Musashino-shi, Tokyo
  - Tokyo Rosai Hospital, Ōta-ku, Tokyo
  - Nissan Tamagawa Hospital, Setagaya-ku, Tokyo
  - Sanin Rosai Hospital, Yonago-shi, Tottori
  - Nihonkai General Hospital, Sakata-shi, Yamagata

IPD SHARING:
Plan to Share IPD: No